CLINICAL TRIAL: NCT03102138
Title: Long Term, Open-Label, Safety Follow Up Study Following Transplantation of Pf-05206388 (Human Embryonic Stem Cell Derived Retinal Pigment Epithelium (RPE)) in Subjects with Acute Wet Age Related Macular Degeneration and Recent Rapid Vision Decline
Brief Title: Retinal Pigment Epithelium Safety Study for Patients in B4711001
Status: Active, not recruiting | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DACL1013; 2015-002267-42 (EudraCT Number)
Record Dates: First submitted 2016-09-22; First posted 2017-04-05 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observation: subjects treated in B4711001 with PF-05206388 will be assessed

SUMMARY:
This is a safety follow-up study. Patients enrolled in B4711001 will be followed for a further 4 years with regular visits to assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Previous participation in Protocol B4711001 and received treatment with PF-05206388.
* Subjects who are willing and able to comply with scheduled visits, and study procedures.

Exclusion Criteria:

* there are no exclusion criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AMD treated in main study
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of serious adverse events and ocular adverse events | 4 years
  incidence of serious adverse events and ocular adverse events will be monitored

SECONDARY OUTCOMES:
Change from baseline (pre-implantation) in ETDRS (Early Treatment of Diabetic Retinopathy Study) best corrected visual acuity (BCVA) | 4 years
  Change from baseline (pre-implantation) in ETDRS (Early Treatment of Diabetic Retinopathy Study) best corrected visual acuity (BCVA). The Proportion of subjects with an improvement of 15 letters or more at all timepoints will be assessed
Mean ETDRS BCVA and change from baseline (pre-implantation) at all timepoints. | 4 years
  Mean ETDRS BCVA and change from baseline (pre-implantation) at all timepoints will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon da Cruz, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B4711005